CLINICAL TRIAL: NCT06609239
Title: An Open Label Extension Study to Evaluate the Long-term Safety and Efficacy of Subcutaneous Lunsekimig in Adult Participants With Asthma Who Participated in Study DRI16762 or ACT18301
Brief Title: Long-term Safety and Efficacy Evaluation of Lunsekimig (SAR443765) in Adult Participants With Asthma.
Acronym: AIRPHRODITE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS17231; 2025-522896-27 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lunsekimig (Experimental): Participants will receive a subcutaneous injection of lunsekimig according to established dosing interval
  Interventions: Drug: Lunsekimig

INTERVENTIONS:
Drug: Lunsekimig — * Pharmaceutical form: Solution for injection in vial
  * Route of administration: Subcutaneous injection
  Other Names: SAR443765

SUMMARY:
This is a phase 2, open-label extension study to evaluate the long-term safety and efficacy of lunsekimig in adult participants with asthma who have previously completed the parent studies. After completion of the parent study, eligible participants will be offered the opportunity to participate in the long-term extension (LTE) study with lunsekimig.

The study duration will be up to 100 weeks with a treatment duration being up to 96 weeks.

DETAILED DESCRIPTION:
Enter Intervention Groups

ELIGIBILITY:
Inclusion Criteria:

1. Participants who completed the 48-week treatment period of Study DRI16762 or ACT18301, including the EOT visit, as per protocol
2. Participants with stable background therapy with moderate or high-dose ICS in combination with the following controller medications, as maintained during the respective parent study in which they have participated:

   * For Study DRI16762: At least 1 and no more than 2 additional controllers (eg, LABA, LAMA, LTRA, or methylxanthines) with or without oral prednisone
   * For Study ACT18301: LABA with or without LTRA
3. Participants who are able and willing to participate in the open-label extension study, and to comply with requested study visits and procedures
4. Contraception for male and female participants

   For female participants:
   * must agree to use contraception/barrier
   * not pregnant or breast feeding
   * no eggs donation or cryopreserving eggs

   For male participants:
   * No sperm donation or cryopreserving sperm
5. Capable of giving signed informed consent

Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

1. Participant who developed a new medical condition or a change in status of an established medical condition or requires a new treatment or medication prior to enrollment that, per Investigator's medical judgement would adversely affect participation of the participant in this study or would require permanent lunsekimig discontinuation, or participants potentially at risk of noncompliance to study procedures
2. Participant who was diagnosed with a new pulmonary disease which may impair lung function
3. Current smoker or active vaping of any products and/or marijuana smoking
4. Prescription drug or substance abuse, including alcohol, considered significant by the Investigator
5. History of hypersensitivity or allergy to lunsekimig or to any of the excipients used in the presentation or in preparation for administration of lunsekimig, or other allergy that, in the opinion of the Investigator, contraindicates participation in the study
6. Participants who are receiving prohibited concomitant medications
7. Participants who, during their participation in the parent study, developed an AE or an SAE deemed related to lunsekimig, which in the opinion of the Investigator could indicate that continued treatment with lunsekimig may present an unreasonable risk for the participant
8. Concurrent participation in any other clinical study, including non-interventional studies
9. Individuals accommodated in an institution because of regulatory or legal order; prisoners or participants who are legally institutionalized
10. Participants are employees of the investigative site or other individuals directly involved in the conduct of the study, or immediate family members of such individuals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2031-01-20 (Estimated); Study Completion 2031-01-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants having any treatmentemergent adverse event (TEAE), including adverse events of special interest (AESI), and serious adverse event (SAE) | From study baseline to week 100

SECONDARY OUTCOMES:
Annualized rate of asthma exacerbation events | From study baseline to week 48
Annualized rate of asthma exacerbation events | From study baseline to week 96
Change from parent study baseline in prebronchodilator (BD) forced expiratory volume in 1 second (FEV1) | From parent study baseline to week 48
Change from parent study baseline in pre bronchodilator (BD) FEV1 | From parent study baseline to week 96
Change from parent study baseline in Asthma Control Questionnaire5 (ACQ-5) score | From parent study baseline to week 48
  The ACQ-5 is a questionnaire that measures the adequacy of asthma control and any changes in asthma control that may occur spontaneously or as a result of treatment. The ACQ-5 has five questions on the asthma symptoms and patients are asked to recall how their asthma has been during the previous week and to respond on a 7-point scale for each question (0 = no impairment, 6 = maximum impairment). The ACQ-5 score is the mean of the 5 questions and, therefore, between 0 (totally controlled) and 6 (severely uncontrolled). A high score indicates low asthma control.
Change from parent study baseline in Asthma Control Questionnaire 5 (ACQ-5) score | From parent study baseline to week 96
Proportion of participants with ≥0.5-point reduction in each score as compared to parent study baseline score | From parent study baseline to week 48
  Defined as ACQ-5 responder analysis
Proportion of participants with ≥0.5-point reduction in each score as compared to parent study baseline score | From parent study baseline to week 96
  Defined as ACQ-5 responder analysis
Change from parent study baseline in Asthma Quality of Life Questionnaire Standardized Activites for 12 years and older (AQLQ[S] +12) domain and total scores | From parent study baseline to week 48
  The AQLQ(S) + 12 was designed as a self-administered patient reported outcome to measure the functional impairments that are most troublesome to adolescents and adults ≥12 years of age as a result of their asthma. The instrument is comprised of 32 items, each rated on a 7-point Likert scales from 1 to 7. Higher scores indicate better quality of life.
Change from parent study baseline in Asthma Quality of Life Questionnaire Standardized Activities for 12 years and older (AQLQ[S] +12) domain and total scores | From parent study baseline to week 96
Serum lunsekimig concentrations | From study baseline to week 100
Incidence and titer of anti-drug antibodies (ADA) against lunsekimig | From study baseline to week 100

CONTACTS AND LOCATIONS:
Locations (114):
- United States (22):
  - Allianz Research Institute - Aurora- Site Number : 8400026, Aurora, Colorado
  - Western States Clinical Research- Site Number : 8400014, Wheat Ridge, Colorado
  - Helix Biomedics- Site Number : 8400114, Boynton Beach, Florida
  - Beautiful Minds Clinical Research Center- Site Number : 8400049, Cutler Bay, Florida
  - Qway Research - Hialeah- Site Number : 8400015, Hialeah, Florida
  - Clintex Research Group - Miami - Southwest 27th Avenue- Site Number : 8400048, Miami, Florida
  - High Quality Research- Site Number : 8400039, Miami, Florida
  - Innovations Biotech- Site Number : 8400040, Miami, Florida
  - New Access Medical Center- Site Number : 8400043, Miami, Florida
  - Deluxe Health Center- Site Number : 8400045, Miami Lakes, Florida
  - Windom Allergy, Asthma and Sinus Specialists- Site Number : 8400019, Sarasota, Florida
  - University of Michigan Health System - Ann Arbor- Site Number : 8400004, Ann Arbor, Michigan
  - Midwest Clinical Research Center - St. Louis- Site Number : 8400006, St Louis, Missouri
  - Tryon Medical Partners - Charlotte - Piedmont Row Drive South- Site Number : 8400029, Charlotte, North Carolina
  - Asthma & Allergy Center - Toledo- Site Number : 8400017, Toledo, Ohio
  - OK Clinical Research- Site Number : 8400021, Edmond, Oklahoma
  - Allergy & Clinical Immunology Associates Pittsburgh- Site Number : 8400007, Pittsburgh, Pennsylvania
  - Orion Clinical Research- Site Number : 8400001, Austin, Texas
  - South Texas Medical Research Institute - TTS Research- Site Number : 8400010, Boerne, Texas
  - Baylor University Medical Center- Site Number : 8400002, Dallas, Texas
  - Western Sky Medical Research- Site Number : 8400023, El Paso, Texas
  - Metroplex Pulmonary and Sleep Center- Site Number : 8400022, McKinney, Texas
- Argentina (10):
  - Investigational Site Number : 0320007, Berazategui, Buenos Aires
  - Investigational Site Number : 0320003, La Plata, Buenos Aires
  - Investigational Site Number : 0320002, Rosario, Santa Fe Province
  - Investigational Site Number : 0320006, Rosario, Santa Fe Province
  - Investigational Site Number : 0320008, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320005, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320009, Mendoza
  - Investigational Site Number : 0320010, Santa Fe
- Brazil (8):
  - Associacao Proar- Site Number : 0760003, Salvador, Estado de Bahia
  - Universidade Federal de Goias- Site Number : 0760007, Goiânia, Goiás
  - Centro de Estudos em Terapias Inovadoras- Site Number : 0760002, Curitiba, Paraná
  - Instituto de Medicina Integral Professor Fernando Figueira- Site Number : 0760009, Recife, Pernambuco
  - Hospital São Lucas da PUCRS - Porto Alegre - Avenida Ipiranga- Site Number : 0760001, Porto Alegre, Rio Grande do Sul
  - Hospital Dia do Pulmão- Site Number : 0760005, Blumenau, Santa Catarina
  - CCBR / IBPClin - Instituto Brasil de Pesquisa Clínica- Site Number : 0760006, Rio de Janeiro
  - Incor - Instituto do Coracao- Site Number : 0760011, São Paulo
- Canada (3):
  - Investigational Site Number : 1240003, Hamilton, Ontario
  - Investigational Site Number : 1240004, Sherbrooke, Quebec
  - Investigational Site Number : 1240001, Trois-Rivières, Quebec
- Chile (7):
  - Investigational Site Number : 1520001, Talca, Maule Region
  - Investigational Site Number : 1520006, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520008, Quillota, Región de Valparaíso
  - Investigational Site Number : 1520011, Viña del Mar, Región de Valparaíso
- China (16):
  - Investigational Site Number : 1560011, Beijing
  - Investigational Site Number : 1560010, Changchun
  - Investigational Site Number : 1560017, Changsha
  - Investigational Site Number : 1560009, Guangzhou
  - Investigational Site Number : 1560001, Guangzhou
  - Investigational Site Number : 1560006, Hefei
  - Investigational Site Number : 1560014, Hohhot
  - Investigational Site Number : 1560007, Nanchang
  - Investigational Site Number : 1560002, Pingxiang
  - Investigational Site Number : 1560013, Shanghai
  - Investigational Site Number : 1560015, Shenyang
  - Investigational Site Number : 1560005, Wenzhou
  - Investigational Site Number : 1560003, Wuhan
  - Investigational Site Number : 1560004, Xuzhou
  - Investigational Site Number : 1560016, Yangzhou
  - Investigational Site Number : 1560012, Zhanjiang
- India (5):
  - Investigational Site Number : 3560009, Hyderabad
  - Investigational Site Number : 3560008, Kanpur
  - Investigational Site Number : 3560007, Kozhikode
  - Investigational Site Number : 3560001, Nagpur
  - Investigational Site Number : 3560004, Pune
- Israel (8):
  - Investigational Site Number : 3760006, Ashkelon
  - Investigational Site Number : 3760001, Haifa
  - Investigational Site Number : 3760008, Haifa
  - Investigational Site Number : 3760003, Jerusalem
  - Investigational Site Number : 3760002, Jerusalem
  - Investigational Site Number : 3760010, Petah Tikva
  - Investigational Site Number : 3760004, Rehovot
  - Investigational Site Number : 3760007, Tel Aviv
- Japan (8):
  - Investigational Site Number : 3920002, Sakaidechō, Kagawa-ken
  - Brigham & Women's Hospital- Site Number : 8400034, Joso-Shi, Massachusetts
  - Investigational Site Number : 3920011, Chūō, Tokyo
  - Investigational Site Number : 3920005, Ube, Yamaguchi
  - Investigational Site Number : 3920008, Fukushima
  - Investigational Site Number : 3920006, Kyoto
  - Investigational Site Number : 3920009, Kyoto
  - Investigational Site Number : 3920012, Miyazaki
- Mexico (6):
  - Investigational Site Number : 4840004, Monterrey, Nuevo León
  - Investigational Site Number : 4840005, San Juan del Río, Querétaro
  - Investigational Site Number : 4840007, Mérida, Yucatán
  - Investigational Site Number : 4840002, Chihuahua City
  - Investigational Site Number : 4840003, Durango
  - Investigational Site Number : 4840008, Veracruz
- South Africa (6):
  - Investigational Site Number : 7100004, Benoni
  - Investigational Site Number : 7100005, Benoni
  - Investigational Site Number : 7100003, Cape Town
  - Investigational Site Number : 7100002, Cape Town
  - Investigational Site Number : 7100001, Durban
  - Investigational Site Number : 7100006, Pretoria
- South Korea (5):
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100006, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100005, Seoul, Seoul-teukbyeolsi
- Turkey (Türkiye) (6):
  - Investigational Site Number : 7920006, Bursa
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920003, Istanbul
  - Investigational Site Number : 7920005, İzmit
  - Investigational Site Number : 7920007, Kayseri
  - Investigational Site Number : 7920001, Mersin
- United Kingdom (4):
  - Investigational Site Number : 8260001, Cambridge, Cambridgeshire
  - Investigational Site Number : 8260004, Glasgow, Glasgow City
  - Investigational Site Number : 8260005, Chertsey, Surrey
  - Investigational Site Number : 8260008, Bradford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LTS17231 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26128&tenant=MT_SNY_9011